CLINICAL TRIAL: NCT03916640
Title: A Trial to Investigate Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of a Co-formulation of an Insulin Analog and Pramlintide in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Trial to Assess a Co-formulation of an Insulin Analog and Pramlintide in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CT034-ADO09
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — pramlintide; Insulin, Regular, Human; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Co-formulation of insulin analog and pramlintide (ADO09) (Experimental): Subcutaneous injection of ADO09 formulation + injection of placebo (0.9% NaCl) to ensure double dummy.
  Interventions: Drug: ADO09 formulation; Drug: Placebo
- Humulin® + Symlin® (Active Comparator): Simultaneous, separate subcutaneous injections of human insulin and pramlintide.
  Interventions: Drug: Symlin®; Drug: Humulin®
- Humalog® (Active Comparator): Subcutaneous injection of insulin lispro + injection of placebo (0.9% NaCl) to ensure double dummy.
  Interventions: Drug: Placebo; Drug: Humalog®

INTERVENTIONS:
Drug: ADO09 formulation — Subcutaneous injection of ADO09 formulation
  Arms: Co-formulation of insulin analog and pramlintide (ADO09)
Drug: Placebo — Subcutaneous injection of 0.9% NaCl
  Arms: Co-formulation of insulin analog and pramlintide (ADO09); Humalog®
Drug: Symlin® — Subcutaneous injection of pramlintide
  Arms: Humulin® + Symlin®
Drug: Humulin® — Subcutaneous injection of human insulin
  Arms: Humulin® + Symlin®
Drug: Humalog® — Subcutaneous injection of insulin lispro
  Arms: Humalog®

SUMMARY:
This trial is a monocentric, randomised, double-blind, active comparator, controlled, 3-period cross-over trial.

DETAILED DESCRIPTION:
In this monocentric, randomised, double-blind, active comparator, controlled, cross-over trial, each patient will be randomly allocated to a sequence of three treatments: one single dose of the co-formulation of insulin analog and pramlintide (also called ADO09), simultaneous separate injections of pramlintide and human insulin and one single dose of insulin lispro. To keep the blinding in this trial, a placebo injection will be given in addition to the ADO09 formulation and insulin lispro dose for a total of 2 injections per dosing visit. During each visit, meal test procedures will be performed and subjects will stay at the clinical centre until post-dose follow-up period has been terminated. IMP administration will be done subcutaneously immediately prior to test meal intake.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus (as diagnosed clinically) ≥ 12 months
* Treated with multiple daily injection ≥ 12 months
* Treated with insulin glargine U100 or U300 or insulin detemir at screening
* Fasting C-peptide ≤ 0.30 nmol/L
* BMI: 18.5-28.0 kg/m² (both inclusive)

Exclusion Criteria:

* Known or suspected hypersensitivity to IMPs, paracetamol or related products
* Type 2 Diabetes Mellitus
* Clinically significant abnormal haematology, biochemistry or urinalysis screening test, as judged by the investigator considering the underlying disease
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea), as judged by the investigator
* Known slowing of gastric emptying, including gastroparesis and or gastrointestinal surgery that in the opinion of the investigator, might change gastrointestinal motility and food absorption
* Intake of medication known to affect gastrointestinal motility, including but not limited to erythromycin, metoclopramide, cisapride, cholestyramine or colestipol within 4 weeks before screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
CmaxPram | From 0 to 8 hours
  Maximum pramlintide concentration
AUCPram 0-8h | From 0 to 8 hours
  Area under the pramlintide concentration-time curve from 0-8 hours after IMP administration
CmaxIns | From 0 to 8 hours
  Maximum insulin analog concentration
AUCIns 0-8h | From 0 to 8 hours
  Area under the insulin analog concentration-time curve from 0-8 hours after IMP administration

SECONDARY OUTCOMES:
Pharmacokinetics of pramlintide | From 0 to 8 hours
  Area under the pramlintide concentration-time curve
Pharmacokinetics of insulins | From 0 to 8 hours
  Area under the insulins concentration-time curve
Glucose pharmacodynamics | From 0 to 8 hours
  Area under the blood glucose concentration-time curve
Safety and tolerability (Adverse Events recording) | From 0 to 8 hours
  Number of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany